CLINICAL TRIAL: NCT02627235
Title: The Deep South IVR-based Active Lifestyle (DIAL) Study
Brief Title: The Deep South IVR-based Active Lifestyle Study
Acronym: DIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dorothy Pekmezi, PhD, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: X131203002; 1R03CA177538 (NIH)
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Physical Activity
Keywords: Physical Activity; Cancer Prevention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DIAL Intervention (Experimental): The physical activity intervention emphasizes behavioral strategies for increasing activity levels (i.e., goal-setting, self-monitoring, problem-solving barriers, increasing social support, rewarding oneself for meeting physical activity goals), and includes daily IVR-system call feedback and monthly graphic-based feedback delivered in the mail. In addition, social support, outcome expectations and perceived physical activity enjoyment variables will be assessed at baseline, 30, 60, and 90 days. Responses will be used to select appropriate tailored feedback modules.
  Interventions: Behavioral: DIAL
- Wait List Control (Active Comparator): Access to the intervention 12 weeks following baseline assessment.
  Interventions: Behavioral: Wait List Control

INTERVENTIONS:
Behavioral: DIAL — The physical activity intervention is based on Social Cognitive Theory and includes feedback on physical activity progress via IVR system and monthly graphic-based feedback letters delivered in the mail. Messages will encourage incremental increases until national PA guidelines are reached and provide specific information on cancer risk reduction.
  Arms: DIAL Intervention
Behavioral: Wait List Control — Access to DIAL intervention 12 weeks following baseline assessment.
  Arms: Wait List Control

SUMMARY:
This pilot study represents an initial foray into delivering an Individual Voice Response-based (IVR) physical activity intervention for cancer risk among sedentary adults in the Deep South.

DETAILED DESCRIPTION:
60 participants will receive the DIAL intervention or Wait List Control. While main outcomes are focused on feasibility and acceptability, physical activity, fitness, and body weight and composition data will be collected and measured at baselines and 12-weeks.

DIAL Intervention: The physical activity intervention is based on Social Cognitive Theory and emphasizes behavioral strategies for increasing activity levels (i.e., goal setting, self-monitoring, problem solving barriers, increasing social support, rewarding oneself for meeting physical activity goals) and includes daily activity reporting via an Individual Voice Response (IVR) system that allows computer-assisted interaction with participants by telephone. Computer expert system feedback on physical activity progress will be based on participants' reported daily step counts and >moderate intensity PA . In addition to IVR system feedback, participants will receive monthly graphic-based feedback letters delivered by mail. Messages will encourage incremental increases until national PA guidelines are reached and provide specific information on cancer risk reduction ("In the past 7 days, you called the DIAL study line all 7 days and reported engaging in 80 minutes of moderate intensity PA. The national guidelines call for >150 min/week of moderate intensity PA so you are well on your way. Keep up the good work. Make small increases in PA each week until you reach that goal. Remember: 30-60 min/day of moderate-vigorous intensity PA may significantly lower your risk of breast and colon cancer").

To improve self-efficacy, social support, outcome expectations, and perceived enjoyment, we will assess these variables at baseline, 30, 60, and 90 days. Responses will be used to select appropriate tailored feedback modules (for low self-efficacy score, "You do not seem confident about your ability to exercise. Often trying to fit in some PA on top of the demands of work and family can be a challenge. Try making time for a 10 minute walk 1-2 days this week. It will help build confidence about your ability to fit PA into your lifestyle.") Finally, participants will receive access to problem solving modules, addressing PA barriers identified by the community during formative research (lack of time, negative outcome expectations, enjoyment, social support, see table below). Module options will be rotated and constantly updated to keep participants engaged.

Wait List Control Condition: Will receive the intervention after 12 weeks following baseline assessments.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older
* Underactive (<60 min/week moderate PA)
* Able to speak/read English
* Willing to be assigned to either condition
* Access to a telephone
* Not planning to move from the area in the next 4 months
* Healthy (BMI 18.5-45; No history of heart disease, myocardial infarction, angina, stroke, or orthopedic conditions which limit mobility, or any serious medical condition that would make physical activity unsafe; no psychiatric hospitalization in past 3 years).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-07; Primary Completion 2017-06 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Consumer Satisfaction Survey | 3 months
  Satisfaction with IVR-based system intervention

SECONDARY OUTCOMES:
7 Day Physical Activity Recall | Baseline and 3 months
  minutes/week of moderate intensity or greater physical activity
6 Minute Walk Test | Baseline and 3 months
  meters walked in 6 minutes
body mass index | Baseline and 3 months
  kg/m^2
waist circumference | Baseline and 3 months
  cm
body impedance analyses | Baseline and 3 months
  % body fat
Social Support for exercise scale | Baseline, 1 month, 2 months, and 3 months
  range=0-65 for both friends and family subscales, with higher scores indicating more social support
Outcome expectations scale | Baseline, 1 month, 2 months, and 3 months
  range= 1-5, with higher scores representing more outcome expectations
Physical Activity Enjoyment scale | Baseline, 1 month, 2 months, and 3 months
  range=18-126, with higher scores indicating more enjoyment
Self -Efficacy for Exercise Measure | Baseline, 1 month, 2 months, and 3 months
  range= 1-5, with higher scores representing more self-efficacy
Accelerometers | Baseline and 3 months
  minutes/week of moderate intensity or greater physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Dori Pekmezi, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No